CLINICAL TRIAL: NCT05912933
Title: Evaluation of Incidence of Myelosuppression (Grade 4 Neutropenia) in Breast Cancer Patients With Mild, Moderate or Severe Hepatic Impairment Treated With Palbociclib Compared to Patients With Reserved Hepatic Function in the Post-marketing Setting: Cohort Study Using the Medical Information Database Network (MID-NET) Database
Brief Title: A Study to Learn About the Relationship Between Hepatic Impairment and Myelosuppression (Decreased Bone Marrow Function) in Breast Cancer Patients Treated With the Study Medicine Palbociclib (Pal-bow-sai-klib)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481116
Record Dates: First submitted 2023-06-11; First posted 2023-06-22 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: Safety; database study in Japan; Ibrance; Palbociclib; hormone receptor-positive (HR+)/human epidermal growth factor receptor 2-negative (HER2-); inoperable or recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- Cohort: New users of palbociclib for inoperable or recurrent breast cancer divided into 4 groups based on severity levels of hepatic impairment

SUMMARY:
The purpose of this study is to evaluate incidence of grade 4 neutropenia in patients who have hepatic impairment and use the study medicine Palbociclib.

This study is seeking participants:

* treated with the study medicine Palbociclib
* having any breast cancer records in same month as the index date (the first prescription date)
* having prescription records of palbociclib from 20 December 2016 to 29 February 2024

The study design is a cohort study. This study design uses de-identified patient data from a hospital based electronic medical record and claim database in Japan.

One of the important side effects of taking Palbociclib is neutropenia (decreased count of neutrophils - a type of white blood cell). In this study, the relationship between neutropenia caused by Palbociclib and hepatic impairment was studied after it was released to the market. To do that, the study gathered details of breast cancer patients newly treated with Palbociclib from 23 hospitals and 10 medical institutes across Japan.

The below patient details were collected:

* dose of Palbociclib
* other medicines prescribed for cancer
* age
* gender
* past information on cancer treatments
* laboratory findings at baseline

The result was based on the neutrophil count collected from the laboratory data. Around 1300 patients newly treated with Palbociclib for breast cancer was calculated by the medical information database network (MID-NET) in 6 years from 15 December 2017.

ELIGIBILITY:
Inclusion Criteria:

* Having prescription records of palbociclib from 15 December 2017 to 29 February 2024.
* Having any breast cancer records in same month as the first prescription date.
* Having laboratory tests and visit records (SS-MIX2) on or before 180 days prior to the first prescription date
* Having SS-MIX2 hospital-visit records within 180 days before the first prescription date

Exclusion Criteria:

* Having an absolute neutrophil count (ANC) less than the threshold value for grade 4 neutropenia within 30 days of the first prescription of palbociclib
* Having any records of anti-HER2 medication

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Breast cancer patients treated with Palbociclib
Sampling Method: Probability Sample
Enrollment: 733 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants With/Without Hepatic Impairment for Grade 4 Neutropenia in New Users of Palbociclib | 20 Dec 2016 through 29 Feb 2024
  Grade 4 neutropenia, as the outcome of this study, will be defined as an ANC of less than 0.5 × 10^9 cells/L or less than 500 cells/mL during the "on-treatment" period.

SECONDARY OUTCOMES:
Number of Participants With/Without Hepatic Impairment for Grade 3-4 Neutropenia in New Users of Palbociclib | 20 Dec 2016 through 29 Feb 2024
  Grade 3-4 neutropenia, as the outcome of this study, will be defined as an ANC of less than 1.0 × 10^9 cells/L or less than 500 cells/mL during the "on-treatment" period.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.